CLINICAL TRIAL: NCT05094232
Title: Epidemiologic Evolution of Coeliac Disease in Spain and Risk Factors Influencing Disease Prevalence
Brief Title: Coeliac Disease in Spain: Determination of Disease Prevalence and Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: EHD20PI01
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies have showed that Coeliac Disease (CD) prevalence is significantly higher in children compared with adults. The largest epidemiologic study carried out in Spain to date (n=4230) reported a higher CD prevalence in children (1:71) than in adults (1:357) during 2004-2007. To study whether this difference was due to environmental factors influencing infancy or the development of gluten tolerance with age, a natural history study in pediatric age was initiated in 2013. Unexpectedly, the prevalence in children of 1-2 years of age was lower (1:135) than the previously reported in 2004-2007 for that age group (1:25). During follow-up, 1/3 of the asymptomatic cases showed reversion of the intestinal lesion and/or negativization of CD serological markers while continuing on a gluten-containing diet. Therefore, the development of gluten tolerance seems to have a major effect in age-related differences in CD prevalence. However, gluten tolerance phenomenon does not explain the differences found between the 2013-2019 and the 2004-2007 cohorts, suggesting that environmental factors may contribute as well. Apart from genetic factors, several environmental factors are believed to influence disease appearance, such as the time that gluten is introduced to the diet, viral infections, type of birth, antibiotic treatments, etc. Therefore, development of tolerance and environmental factors seem to equally play an important role in age-related differences in CD prevalence. However, more data is needed in order to know how environmental factors influence disease prevalence in Spain. Also, the previous studies carried in Spain were performed in specific geographical areas: Asturias, Basque Country and Catalonia using slightly different methodology and focused on different age groups, thus making results comparison and global extrapolation challenging.

In this study, the investigators aim to determine global CD prevalence in Spain during 2020-2021 and: 1) compare it with the results obtained in previous studies; and 2) identify whether there are any differences associated with age, environmental factors and/or geographical area. For this purpose: a) participants are recruited based on the reference population regarding age and gender; b) recruitment is done in 5 different geographical areas in Spain: Andalusia, Asturias, Basque Country, Catalonia and Madrid; c) relevant clinical, social and environmental data is collected and d) serologic screening (anti-tissue transglutaminase (tTG) - Immunoglobulin A (IgA) antibodies detection in blood serum) with histological confirmation (small-intestinal biopsy) is used to detect CD cases and determine disease prevalence.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 to ≥80 years old

Exclusion Criteria:

* Heart failure or unstable ischemic cardiopathy
* Chronic obstructive pulmonary disease or respiratory insufficiency
* Coagulopathy
* Diabetes mellitus type II with vascular complications
* Hepatic cirrhosis
* Kidney failure (Creatinine >1.5 mg/dL o glomerular filtration <30 ml /min)
* Active neoplasm
* Pregnancy
* Gluten-free diet without CD diagnosis

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants are selected from ambulatory minor surgery departments of the pediatric and general tertiary referral hospitals in Spain. Regarding age and sex, inclusion is done reproducing the reference population of each participating Spanish regions (according to data from the Spanish Statistics Institute).
Sampling Method: Non-Probability Sample
Enrollment: 5255 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
tissue transglutaminase IgA antibodies (tTGA) detection in blood serum (serological CD marker) | at the time of recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Singh P, Arora A, Strand TA, Leffler DA, Catassi C, Green PH, Kelly CP, Ahuja V, Makharia GK. Global Prevalence of Celiac Disease: Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2018 Jun;16(6):823-836.e2. doi: 10.1016/j.cgh.2017.06.037. Epub 2018 Mar 16. PMID 29551598
- [Background] Pratesi R, Gandolfi L, Garcia SG, Modelli IC, Lopes de Almeida P, Bocca AL, Catassi C. Prevalence of coeliac disease: unexplained age-related variation in the same population. Scand J Gastroenterol. 2003 Jul;38(7):747-50. doi: 10.1080/00365520310003255. PMID 12889561
- [Background] Beatriz Arau; Meritxell Mariné; Carme Farré; Beatriz Dietl; Roger García-Puig; Laura Martí-Cosconera; Anna Carrasco; Eva Tristán; Teresa Marqués; Víctor Vila; Clàudia Fortuny, Maria Esteve. Història natural de la malaltia celíaca (MC): seguiment longitudinal a llarg termini amb dieta lliure de nens asimptomàtics detectats per cribratge poblacional. Resultats preliminars. XXVII Congrés de la Societat Catalana de Digestologia. Girona: 25-27 de gener de 2018. (Annals de Medicina 2018; Suplements Vol. 101 supl. 1)
- [Background] Myleus A, Ivarsson A, Webb C, Danielsson L, Hernell O, Hogberg L, Karlsson E, Lagerqvist C, Norstrom F, Rosen A, Sandstrom O, Stenhammar L, Stenlund H, Wall S, Carlsson A. Celiac disease revealed in 3% of Swedish 12-year-olds born during an epidemic. J Pediatr Gastroenterol Nutr. 2009 Aug;49(2):170-6. doi: 10.1097/MPG.0b013e31818c52cc. PMID 19516192
- [Background] Szajewska H, Shamir R, Chmielewska A, Piescik-Lech M, Auricchio R, Ivarsson A, Kolacek S, Koletzko S, Korponay-Szabo I, Mearin ML, Ribes-Koninckx C, Troncone R; PREVENTCD Study Group. Systematic review with meta-analysis: early infant feeding and coeliac disease--update 2015. Aliment Pharmacol Ther. 2015 Jun;41(11):1038-54. doi: 10.1111/apt.13163. Epub 2015 Mar 26. PMID 25819114
- [Background] Namatovu F, Lindkvist M, Olsson C, Ivarsson A, Sandstrom O. Season and region of birth as risk factors for coeliac disease a key to the aetiology? Arch Dis Child. 2016 Dec;101(12):1114-1118. doi: 10.1136/archdischild-2015-310122. Epub 2016 Aug 15. PMID 27528621
- [Background] Zanoni G, Navone R, Lunardi C, Tridente G, Bason C, Sivori S, Beri R, Dolcino M, Valletta E, Corrocher R, Puccetti A. In celiac disease, a subset of autoantibodies against transglutaminase binds toll-like receptor 4 and induces activation of monocytes. PLoS Med. 2006 Sep;3(9):e358. doi: 10.1371/journal.pmed.0030358. PMID 16984219
- [Background] Kahrs CR, Chuda K, Tapia G, Stene LC, Marild K, Rasmussen T, Ronningen KS, Lundin KEA, Kramna L, Cinek O, Stordal K. Enterovirus as trigger of coeliac disease: nested case-control study within prospective birth cohort. BMJ. 2019 Feb 13;364:l231. doi: 10.1136/bmj.l231. PMID 30760441
- [Background] Kemppainen KM, Lynch KF, Liu E, Lonnrot M, Simell V, Briese T, Koletzko S, Hagopian W, Rewers M, She JX, Simell O, Toppari J, Ziegler AG, Akolkar B, Krischer JP, Lernmark A, Hyoty H, Triplett EW, Agardh D; TEDDY Study Group. Factors That Increase Risk of Celiac Disease Autoimmunity After a Gastrointestinal Infection in Early Life. Clin Gastroenterol Hepatol. 2017 May;15(5):694-702.e5. doi: 10.1016/j.cgh.2016.10.033. Epub 2016 Nov 10. PMID 27840181
- [Background] Lindfors K, Lin J, Lee HS, Hyoty H, Nykter M, Kurppa K, Liu E, Koletzko S, Rewers M, Hagopian W, Toppari J, Ziegler AG, Akolkar B, Krischer JP, Petrosino JF, Lloyd RE, Agardh D; TEDDY Study Group. Metagenomics of the faecal virome indicate a cumulative effect of enterovirus and gluten amount on the risk of coeliac disease autoimmunity in genetically at risk children: the TEDDY study. Gut. 2020 Aug;69(8):1416-1422. doi: 10.1136/gutjnl-2019-319809. Epub 2019 Nov 19. PMID 31744911
- [Background] Namatovu F, Olsson C, Lindkvist M, Myleus A, Hogberg U, Ivarsson A, Sandstrom O. Maternal and perinatal conditions and the risk of developing celiac disease during childhood. BMC Pediatr. 2016 Jun 8;16:77. doi: 10.1186/s12887-016-0613-y. PMID 27267234
- [Background] Kemppainen KM, Vehik K, Lynch KF, Larsson HE, Canepa RJ, Simell V, Koletzko S, Liu E, Simell OG, Toppari J, Ziegler AG, Rewers MJ, Lernmark A, Hagopian WA, She JX, Akolkar B, Schatz DA, Atkinson MA, Blaser MJ, Krischer JP, Hyoty H, Agardh D, Triplett EW; Environmental Determinants of Diabetes in the Young (TEDDY) Study Group. Association Between Early-Life Antibiotic Use and the Risk of Islet or Celiac Disease Autoimmunity. JAMA Pediatr. 2017 Dec 1;171(12):1217-1225. doi: 10.1001/jamapediatrics.2017.2905. PMID 29052687
- [Background] Dydensborg Sander S, Nybo Andersen AM, Murray JA, Karlstad O, Husby S, Stordal K. Association Between Antibiotics in the First Year of Life and Celiac Disease. Gastroenterology. 2019 Jun;156(8):2217-2229. doi: 10.1053/j.gastro.2019.02.039. Epub 2019 Mar 2. PMID 30836095
- [Background] Riestra S, Fernandez E, Rodrigo L, Garcia S, Ocio G. Prevalence of Coeliac disease in the general population of northern Spain. Strategies of serologic screening. Scand J Gastroenterol. 2000 Apr;35(4):398-402. doi: 10.1080/003655200750023967. PMID 10831263
- [Background] Castano L, Blarduni E, Ortiz L, Nunez J, Bilbao JR, Rica I, Martul P, Vitoria JC. Prospective population screening for celiac disease: high prevalence in the first 3 years of life. J Pediatr Gastroenterol Nutr. 2004 Jul;39(1):80-4. doi: 10.1097/00005176-200407000-00016. PMID 15187786
- [Background] Marine M, Farre C, Alsina M, Vilar P, Cortijo M, Salas A, Fernandez-Banares F, Rosinach M, Santaolalla R, Loras C, Marques T, Cusi V, Hernandez MI, Carrasco A, Ribes J, Viver JM, Esteve M. The prevalence of coeliac disease is significantly higher in children compared with adults. Aliment Pharmacol Ther. 2011 Feb;33(4):477-86. doi: 10.1111/j.1365-2036.2010.04543.x. Epub 2010 Dec 19. PMID 21166832